CLINICAL TRIAL: NCT06439303
Title: Analysis and Evaluation of Smoking Treatment With Cytisine: Retrospective Observational Study
Brief Title: Analysis and Evaluation of Smoking Treatment With Cytisine
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS104/IRE/24
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Moderate or Severe Tobacco Use Disorder
MeSH Terms: conditions — Lymphoma, Follicular; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with moderate or severe tobacco use disorder.: Patients hospitalized at the IRE anti-smoking center, National Cancer Institute "Regina Elena", suffering from moderate or severe tobacco use disorder, who are prescribed pharmacological therapy with Cytisine 1.5 mg.
  Interventions: Drug: Cytisine 1,5 mg

INTERVENTIONS:
Drug: Cytisine 1,5 mg — Administration of Cytisine as monotherapy in the treatment of moderate tobacco use disorder or serious

SUMMARY:
The lack of clinical studies on the use of Cytisine in the treatment of the cessation of smoking, the need to find effective therapeutic alternatives and the opportunity to reduce costs related to the complications of cigarette smoking, represent the main reasons that led to the design of this study.

DETAILED DESCRIPTION:
The study is observational, retrospective and monocentric, and aims to evaluate patients who performed an initial pneumological examination at the Anti-Smoking Center of the National Institute Regina Elena tumors due to smoking cessation in the reference period. To such patients, affected of moderate or severe tobacco use disorder, drug therapy was prescribed with Cytisine 1.5 mg, with the aim of evaluating treatment adherence, efficacy and tolerability of Cytisine as monotherapy in the treatment of moderate or moderate tobacco use disorder serious. Responding patients will be taken into consideration for the study consecutively to the criteria established and pertaining to the Anti-Smoking Center of the National Cancer Institute Regina Elena in the period between 02/01/2023 and 11/30/2023 on first and subsequent visits controls.

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years;
* patients suffering from moderate or severe tobacco use disorder;
* prescription of pharmacological therapy with Cytisine;
* patients returned to the 1st check-up on schedule;

Exclusion Criteria:

* Patients with contraindications to taking Cytisine and partial receptor agonists nicotinic cholinergics;
* Patients undergoing pharmacological or physical treatment for neoplastic pathology;
* Pregnant or breastfeeding women;
* Patients for whom specific information for objective assessments is not available;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have referred to the Anti-smoking Center of the IRE, National Cancer Institute "Regina Elena", and that meet the following criteria.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Therapeutic adherence | 3 months
  Evaluation of adherence to the prescribed drug therapy i.e. Cytisine 1.5 mg

SECONDARY OUTCOMES:
Evaluation of the effectiveness of the therapy. | 3 months
  Evaluation of the effectiveness of the therapy with the achievement of smoking cessation subsequent checks occurred after clinical evaluation and measurement of the monoxide value exhaled carbon.
Evaluation of therapeutic adherence in relation to motivation. | 3 months
  Evaluation of adherence to Cytisine therapy in relation to the patient's motivation measured with the Mondor motivational test.
Assessment of adherence in relation to the dependency score physics. | 3 months
  Evaluation of adherence to Cytisine therapy in relation to the addiction score physical measured with the Nicotine dependence questionnaire or Fagerström test.
Safety and Tolerability assessment. | 3 months
  Safety and Tolerability assessment describing any adverse reactions related to the intake of Cytisine.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy